CLINICAL TRIAL: NCT05954962
Title: Evaluation of the Efficacy of Micronized Natural Progesterone (Seidigestan®) Vs GnRH Antagonist (Astarté®) in the Prevention of LH Peak During Controlled Ovarian Stimulation: a Randomized Clinical Trial.
Brief Title: Efficacy of Micronized Natural Progesterone Vs GnRH Antagonist in the Prevention of LH Peak During Ovarian Stimulation.
Acronym: PRO_NAT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Maria Martinez Moya, Principal Investigator, Instituto Bernabeu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBMR43
Record Dates: First submitted 2023-07-12; First posted 2023-07-20 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: IVF
MeSH Terms: interventions — Progesterone; ganirelix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CONTROL GROUP (Active Comparator): The patient will start to administer: (1) daily subcutaneous injections of gonadotropins on day 1 of ovarian stimulation (2) daily subcutenous injections of ganirelix ("antagonist") on day 5 or 6 of ovarian stimulation. Both medication will be stopped 1-2 days before egg retrieval.
  Interventions: Drug: Ganirelix Acetate
- STUDY GROUP (Experimental): The patient will start to administer: (1) daily subcutaneous injections of gonadotropins on day 1 of ovarian stimulation (2) daily oral capsules of natural micronized progesterone on day 1 of ovarian stimulation. Both medication will be stopped 1-2 days before egg retrieval.
  Interventions: Drug: Progesterone 200 MG

INTERVENTIONS:
Drug: Progesterone 200 MG — The patients in the study group will administer oral natural micronized progesterone capsules from day 1 of ovarian stimulation instead of "antagonist" (ganirelix) subcutaneaous injections from day 5-6 of stimulation.
  Arms: STUDY GROUP
Drug: Ganirelix Acetate — The patients in the control group will administer subcutaneaous injections of ganirelix from day 5-6 of stimulation as per currently used protocol.
  Arms: CONTROL GROUP

SUMMARY:
This study aims to investigate if the use of oral micronized natural progesterone is not inferior to the use of subcutaneous antagonist in preventing LH peak in controlled ovarian stimulation.

DETAILED DESCRIPTION:
The study will aim to include 150 women (egg donors): 75 per group and the principal variable will be the number of retrieved mature (MII) oocytes. Randomized, prospective, controlled, single center, phase IV study.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility for the oocyte donation program at Instituto Bernabeu.
* Age between 18 and 33 years
* BMI >18 and <30
* Overall antral follicle count >8
* Presence of both ovaries
* Ability to participate and comply with the study protocol
* Oral and written comprehension of Spanish
* Having given written consent

Exclusion Criteria:

* Endometriosis at any stage
* Any ovarian tumor whether benign or malignant
* Concurrent participation in another study
* Malabsorptive syndromes that may alter the efficacy of Seidigestan ® such as bariatric surgery, ulcerative colitis or Crohn's disease
* Irregular periods
* Hypogonadotropic hypogonadism
* Having received in the previous two months treatment with ovulation stimulators
* Having previously participated in the present study

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
MII oocytes | Egg collection day (between 8 and 14 days after starting of ovarian stimulation)
  number of mature (MII) oocytes in both stimulations.

SECONDARY OUTCOMES:
Duration | Egg collection day (between 8 and 14 days after starting of ovarian stimulation)
  duration of ovarian stimulation under both protocols.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No
The information collected in the study will always be treated as grouped data and never as individual or personal data, thus maintaining anonymity and confidentiality.

REFERENCES:
- [Background] A double-blind, randomized, dose-finding study to assess the efficacy of the gonadotrophin-releasing hormone antagonist ganirelix (Org 37462) to prevent premature luteinizing hormone surges in women undergoing ovarian stimulation with recombinant follicle stimulating hormone (Puregon). The ganirelix dose-finding study group. Hum Reprod. 1998 Nov;13(11):3023-31. PMID 9853849
- [Background] Balasch J, Creus M, Fabregues F, Carmona F, Casamitjana R, Penarrubia J, Rivera F, Vanrell JA. Hormonal profiles in successful and unsuccessful implantation in IVF-ET after combined GnRH agonist/gonadotropin treatment for superovulation and hCG luteal support. Gynecol Endocrinol. 1995 Mar;9(1):51-8. doi: 10.3109/09513599509160191. PMID 7793300
- [Background] Begueria R, Garcia D, Vassena R, Rodriguez A. Medroxyprogesterone acetate versus ganirelix in oocyte donation: a randomized controlled trial. Hum Reprod. 2019 May 1;34(5):872-880. doi: 10.1093/humrep/dez034. PMID 30927417
- [Background] Castillo JC, Haahr T, Martinez-Moya M, Humaidan P. Gonadotropin-releasing hormone agonist for ovulation trigger - OHSS prevention and use of modified luteal phase support for fresh embryo transfer. Ups J Med Sci. 2020 May;125(2):131-137. doi: 10.1080/03009734.2020.1736696. Epub 2020 May 4. PMID 32366146
- [Background] Fauser BC, Devroey P. Why is the clinical acceptance of gonadotropin-releasing hormone antagonist cotreatment during ovarian hyperstimulation for in vitro fertilization so slow? Fertil Steril. 2005 Jun;83(6):1607-11. doi: 10.1016/j.fertnstert.2005.02.011. PMID 15950626
- [Background] Giles J, Alama P, Gamiz P, Vidal C, Badia P, Pellicer A, Bosch E. Medroxyprogesterone acetate is a useful alternative to a gonadotropin-releasing hormone antagonist in oocyte donation: a randomized, controlled trial. Fertil Steril. 2021 Aug;116(2):404-412. doi: 10.1016/j.fertnstert.2021.02.036. Epub 2021 Apr 2. PMID 33814126
- [Background] Griesinger G, Dawson A, Schultze-Mosgau A, Finas D, Diedrich K, Felberbaum R. Assessment of luteinizing hormone level in the gonadotropin-releasing hormone antagonist protocol. Fertil Steril. 2006 Mar;85(3):791-3. doi: 10.1016/j.fertnstert.2005.08.048. PMID 16500366
- [Background] Guo YC, Chen PY, Li TT, Jia L, Sun P, Zhu WS, Deng CC, Fang C, Liang XY. Different progestin-primed ovarian stimulation protocols in infertile women undergoing in vitro fertilization/intracytoplasmic sperm injection: an analysis of 1188 cycles. Arch Gynecol Obstet. 2019 Apr;299(4):1201-1212. doi: 10.1007/s00404-019-05065-4. Epub 2019 Mar 9. PMID 30852654
- [Background] Kuang Y, Chen Q, Fu Y, Wang Y, Hong Q, Lyu Q, Ai A, Shoham Z. Medroxyprogesterone acetate is an effective oral alternative for preventing premature luteinizing hormone surges in women undergoing controlled ovarian hyperstimulation for in vitro fertilization. Fertil Steril. 2015 Jul;104(1):62-70.e3. doi: 10.1016/j.fertnstert.2015.03.022. Epub 2015 May 5. PMID 25956370
- [Background] Macklon NS, Stouffer RL, Giudice LC, Fauser BC. The science behind 25 years of ovarian stimulation for in vitro fertilization. Endocr Rev. 2006 Apr;27(2):170-207. doi: 10.1210/er.2005-0015. Epub 2006 Jan 24. PMID 16434510
- [Background] Messinis IE, Templeton AA. Endocrine and follicle characteristics of cycles with and without endogenous luteinizing hormone surges during superovulation induction with pulsatile follicle-stimulating hormone. Hum Reprod. 1987 Jan;2(1):11-6. doi: 10.1093/oxfordjournals.humrep.a136481. PMID 3106404
- [Background] Porter RN, Smith W, Craft IL, Abdulwahid NA, Jacobs HS. Induction of ovulation for in-vitro fertilisation using buserelin and gonadotropins. Lancet. 1984 Dec 1;2(8414):1284-5. doi: 10.1016/s0140-6736(84)92840-x. No abstract available. PMID 6150318
- [Background] Yu S, Long H, Chang HY, Liu Y, Gao H, Zhu J, Quan X, Lyu Q, Kuang Y, Ai A. New application of dydrogesterone as a part of a progestin-primed ovarian stimulation protocol for IVF: a randomized controlled trial including 516 first IVF/ICSI cycles. Hum Reprod. 2018 Feb 1;33(2):229-237. doi: 10.1093/humrep/dex367. PMID 29300975
- [Background] Zhu X, Ye H, Fu Y. Duphaston and human menopausal gonadotropin protocol in normally ovulatory women undergoing controlled ovarian hyperstimulation during in vitro fertilization/intracytoplasmic sperm injection treatments in combination with embryo cryopreservation. Fertil Steril. 2017 Sep;108(3):505-512.e2. doi: 10.1016/j.fertnstert.2017.06.017. Epub 2017 Jul 8. PMID 28697910
- [Derived] Martinez-Moya M, Guerrero J, Girela JL, Pitas A, Bernabeu A, Bernabeu R, Castillo JC. Micronized natural progesterone (Seidigestan(R)) vs GnRH antagonists for preventing the LH surge during controlled ovarian stimulation (PRO_NAT study): study protocol of a randomized clinical trial. Front Endocrinol (Lausanne). 2024 Mar 21;15:1350154. doi: 10.3389/fendo.2024.1350154. eCollection 2024. PMID 38577571